CLINICAL TRIAL: NCT01643174
Title: Predictors of Mortality and Morbidity in the Surgical Management of Primary Tumors of the Spine: A Multi-center Retrospective Cohort Study With a Cross-Sectional Survival Check
Brief Title: Predictors of Mortality and Morbidity in the Surgical Management of Primary Tumors of the Spine
Acronym: PT
Status: Completed | Type: Observational
Sponsor: AO Foundation, AO Spine (Other)
Responsible Party: Sponsor
Other Study IDs: PT retro
Record Dates: First submitted 2012-04-17; First posted 2012-07-18 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Spine Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical treatment

SUMMARY:
Within defined groups of primary malignant and benign bone and soft tissue spine tumors, what variables (clinical, diagnostic, therapeutic, and/or demographic) are associated with overall survival?

DETAILED DESCRIPTION:
Primary tumors of the spine are exceedingly rare and therefore the literature has been limited to case series of limited size and significant heterogeneity. These tumors comprise 11% of all Primary Musculoskeletal Tumors and 4.2% of all spine tumors. Of all primary spine tumors only 6% are malignant, but it is the malignant tumors that present the greatest therapeutic challenges. Through this multi-center retrospective cohort study performed at 13 spine oncology referral, data on at least 2.000 patients with specific primary benign and malignant spine tumors will be collected. This will provide power to determine the influence of many previously hypothesized variables on outcome.

The purpose of this study is to determine clinical, imaging and treatment factors that influence patient survival, local recurrence rate, and peri-operative/post-operative morbidity. Most surgical options carry significant morbidity and consume vast resources. In contrast, there is emerging evidence that incomplete or oncologically inappropriate resection increases local recurrence rate and decreases overall survival. These data will be used to refine existing study questions regarding patient outcomes and to develop new study questions that will be assessed in the future using prospectively collected data.

ELIGIBILITY:
Inclusion Criteria:

* Were admitted to one of the participating spine centers with a diagnosis of primary tumor of the spine and were treated surgically.
* At least one follow-up detectable in the medical charts

Exclusion Criteria:

* metastatic tumor of the spine
* primary spinal cord tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective chart review and selection
Sampling Method: Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2012-02; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
overall survival | Average of 10 years

SECONDARY OUTCOMES:
local recurrence | Average of 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Fisher, Vancouver, Canada

REFERENCES:
- [Derived] Disch AC, Boriani S, Luzzati A, Rhines LD, Fisher CG, Lazary A, Gokaslan ZL, Chou D, Clarke MJ, Fehlings MG, Schaser KD, Germscheid NM, Reynolds JJ, The Ao Spine Knowledge Forum Tumor. Extradural Primary Malignant Spinal Tumors in a Population Younger than 25 Years: An Ambispective International Multicenter Study on Onco-Surgical Outcomes. Cancers (Basel). 2023 Jan 30;15(3):845. doi: 10.3390/cancers15030845. PMID 36765803
- [Derived] Fisher CG, Goldschlager T, Boriani S, Varga PP, Rhines LD, Fehlings MG, Luzzati A, Dekutoski MB, Reynolds JJ, Chou D, Berven SH, Williams RP, Quraishi NA, Bettegowda C, Gokaslan ZL. An evidence-based medicine model for rare and often neglected neoplastic conditions. J Neurosurg Spine. 2014 Nov;21(5):704-10. doi: 10.3171/2014.7.SPINE13954. Epub 2014 Sep 5. PMID 25192373